CLINICAL TRIAL: NCT04415203
Title: Efficacy and Safety of Transcutaneous Auricular Vagus Nerve Stimulation for Frequent Premature Ventricular Complexes: A Randomized Controlled Trial
Brief Title: TAES for FPVCs: a Pragmatic, Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: China Association for Science and Technology (Unknown)
Responsible Party: Principal Investigator, Jiani Wu, Dr, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAESforFPVC
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Premature Ventricular Complexes
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVNS plus usual care (Experimental): TAVNS on Erzhong and Xin (Auricular Acupuncture Point with Vagus nerve distribution); Usual Care: usual medicine treatment for PVCs.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (TAVNS)
- Sham-TAVNS plus usual care (Placebo Comparator): Sham-TAVNS on Erzhong and Xin (Auricular Acupuncture Point); the same acupoints as the treatment group without any current.
  Usual Care: usual medicine treatment for PVCs.
  Interventions: Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham-TAVNS)

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (TAVNS) — Patients in TAVNS group will receive TAVNS and usual care. TAVNS will be performed on Erzhong and Xin (Auricular Acupuncture Point with vagus nerve distribution) for 6 weeks by using the Huato type SDZ-V stimulator; Usual Care: usual medicine treatment for PVCs.
  Arms: TAVNS plus usual care
Device: Sham Transcutaneous Auricular Vagus Nerve Stimulation (Sham-TAVNS) — Patients in sham-TAVNS group will receive sham-TAVNS and usual care. Sham-TAVNS will be also performed on Erzhong and Xin (Auricular Acupuncture Point with vegas nerve stimulation) for 6 weeks by using a special Huato type SDZ-V stimulator. We cut the inner electric wire of the stimulator; therefore, there is no current output. Usual Care: usual medicine treatment for PVCs.
  Arms: Sham-TAVNS plus usual care

SUMMARY:
This prospective, randomized controlled trial aims to evaluate the efficacy and safety of Transcutaneous Auricular Vagus Nerve Stimulation (TAVNS) for patients with frequent premature ventricular coomplexes (FPVCs). Ninety participants will be randomized to TAVNS group and sham-TAVNS group with the ratio of 1:1. They will receive TAVNS plus usual care or sham-TAVNS plus usual care for 6 weeks, and then be followed up for 12 weeks after the treatment. The primary outcome was the proportion of participants with a 50% decrease of the 24 hour (24h) premature ventricular complexes (PVCs) after 6-week treatment. Secondary outcomes include the proportion of participants with a 75% decrease of the 24h-PVCs; the decrease from baseline of 24h-PVCs, total 24h-heartbeat, and the frequency of supraventricular arrhythmia; the score change from baseline in PVCs-related symptoms; the score change from baseline in SAS and SDS. Subgroup analyses will be performed in age, gender, and the severity of PVCs. Safety assessment will be documented during the whole trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as frequent premature ventricular contractions;
* 2 ≤ Lown level ≤ 4A;
* 18 ≤ age ≤ 75;
* Volunteered to participant

Exclusion Criteria:

* Severe valvular disease, congenital heart disease, pericardial disease, hypertrophic cardiomyopathy, unstable angina pectoris, acute myocardial infarction, myocarditis, aneurysm, congestive heart failure decompensation period (NYHA grade III or VI), cardiogenic shock, cerebrovascular disease, hematopoietic system disease, severe mental disease;
* Bradycardia, including pathologic sinus node syndrome, degree II or greater atrioventricular block;
* Those who have already had pacemaker or percutaneous coronary intervention, or who plan to have pacemaker or percutaneous coronary intervention;
* Pregnant or lactating women;
* Local sensory deficit, or allergic to current;
* May be allergic to percutaneous patches；
* Blood pressure ≤ 90/60 mmHg;
* Those who have participated in other clinical trials within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the proportion of participants with a 50% decrease of PVCs from baseline | week 6
  The PVCs will be assessed by a 24-hour Holter monitoring. The investigators will calculate the decrease of PVCs between baseline and week 6 (at the end of the treatment), then we will obtain the proportion of patients with a 50% decrease.

SECONDARY OUTCOMES:
the proportion of participants with a 50% decrease of PVCs from baseline | week 18
  The PVCs will be assessed by a 24-hour Holter monitoring. The investigators will calculate the decrease of PVCs between baseline and week 18 (at the end of the follow-up period), then we will obtain the proportion of patients with a 50% decrease.
the proportion of participants with a 75% decrease of PVCs from baseline | week 6, week 18
  The PVCs will be assessed by a 24-hour Holter monitoring. The investigators will calculate the decrease of PVCs between baseline and week 6/18, then we will obtain the proportion of patients with a 75% decrease.
the change from baseline in PVCs | week 6, week 18
  The PVCs will be assessed by a 24-hour Holter monitoring. The investigators will calculate the decrease of PVCs between baseline and week 6/18.
the change from baseline in total cardiac impulse | week 6, week 18
  The total cardiac impulse will be assessed by a 24-hour Holter monitoring. The investigators will calculate the change of total cardiac impulse between baseline and week 6/18.
the change from baseline in supraventricular premature contractions | week 6, week 18
  The change from baseline in supraventricular premature contractions will be assessed by a 24-hour Holter monitoring. The investigators will calculate the change of supraventricular premature contractions between baseline and week 6/18.
the score change from baseline in the symptom of palpitation | week 6, week 18.
  The symptom of palpitation will be assessed by a 10-scale VAS from 0 to 10, a higher score indicates a more severe symptom of palpitation. The investigators will calculate the score change of palpitation between baseline and week 6/18.
the score change from baseline in the symptom of chest tightness | week 6, week 18.
  The symptom of chest tightness will be assessed by a 10-scale VAS from 0 to 10, a higher score indicates a more severe symptom of chest tightness. The investigators will calculate the score change of chest tightness between baseline and week 6/18.
the score change from baseline in the symptom of dizziness | week 6, week 18.
  The symptom of dizziness will be assessed by a 10-scale VAS from 0 to 10, a higher score indicates a more severe symptom of dizziness. The investigators will calculate the score change of dizziness between baseline and week 6/18.
the score change from baseline in the symptom of insomnia | week 6, week 18.
  The symptom of insomnia will be assessed by a 10-scale VAS from 0 to 10, a higher score indicates a more severe symptom of insomnia. The investigators will calculate the score change of insomnia between baseline and week 6/18.
the change of the proportion of participants with moderate/severe symptoms of palpitation, chest tightness, dizziness or insomnia from baseline | week 6, week 18.
  The symptom of palpitation/chest tightness/dizziness/insomnia will be assessed by a 10-scale VAS from 0 to 10. Score 4-6 are defined as the moderate level, Score 7-10 are defined as the severe level. The investigators will calculate the change of the proportion of patients with the moderate/severe symptoms between baseline and week 6/18.
the score change from baseline in the SAS | week 6, week 18.
  Self Anxiety Scale (SAS) contains 20 items scored from 25 to 100. Score 50-59 was classified as mild anxiety; Score 60-69 as moderate anxiety, and score ≥ 70 as severe anxiety.
the score change from baseline in the SDS | week 6, week 18.
  Self Depression Scale (SDS) contains 20 items scored from 25 to 100. Score 53-62 was classified as mild depression; Score 63-72 as moderate depression, and score ≥ 73 as severe depression.
the score change from baseline in SF-36 | week 6, week 18.
  The SF-36 questionnaire contains eight scales with two measures: physical and mental health. The physical health includes four scales of physical functioning (PF), role-physical (RF), bodily pain (BP), and general health (GH). The mental health is composed of vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH).
  SF-36 scores from 0 to 100, higher scores indicate better health status.

OTHER OUTCOMES:
subgroup analysis of ages | week 6
  Subgroup analysis will be performed in the primary outcome. The investigators will classify the patients with two subgroups by age: ≤40 years and > 40 years.
subgroup analysis of gender | week 6
  Subgroup analysis will be performed in the primary outcome. The investigators will classify the patients with two subgroups by gender: male and female.
subgroup analysis of the severity of PVCs | week 6
  Subgroup analysis will be performed in the primary outcome. The investigators will classify the patients with three subgroups by the severity of PVCs through Lown: level 2, level 3, and level 4A
the proportion of participants with adverse events | week 6, week 18
  Safety assessment, The investigators will calculate the adverse events during the whole study.

CONTACTS AND LOCATIONS:
Overall Officials: Jiani Wu, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospita, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu Y, Wei X, Wang L, Yang Y, Xu L, Sun T, Yang L, Cai S, Liu X, Qin Z, Bin L, Sun S, Lu Y, Cui J, Liu Z, Wu J. Efficacy and safety of transcutaneous auricular vagus nerve stimulation for frequent premature ventricular complexes: rationale and design of the TASC-V trial. BMC Complement Med Ther. 2024 Jul 29;24(1):288. doi: 10.1186/s12906-024-04568-1. PMID 39075454